CLINICAL TRIAL: NCT07308093
Title: Effects of Virtual Reality and Proprioceptive Neuromuscular Facilitation on Upper Limb Sensorimotor Control Among Patients With Parkinson's Disease.
Brief Title: Comparative Effects of Virtual Reality and Proprioceptive Neuromuscular Facilitation in Patients With Parkinson's Disease
Acronym: VR PNF RPT PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Prof. Dr. Shoaib Waqas, Dean-0Study Chair, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPT/ERB/33; U1111-1332-3369 (Registry Identifier: Fatima Rehan)
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Sensorimotor Control; Virtual Reality Therapy; Proprioceptive Neuromuscular Facilitation; Upper Limb Rehabilitation; Neuroplasticity
MeSH Terms: conditions — Parkinson Disease | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Not Needed
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants in this group received Virtual Reality (VR)-based training in addition to Routine Physical Therapy (RPT). The VR intervention was delivered using the Oculus Meta Quest 3 headset and consisted of immersive, goal-directed tasks performed three times per week for six weeks, each session lasting 30 minutes at a moderate intensity (RPE 11-13). VR tasks were designed to target specific motor impairments, including pick-and-place tasks for kinetic tremor reduction, tracing tasks to address bradykinesia, and reaching and grasping tasks to improve proprioception. Participants interacted with five virtual balls in a simulated environment, transferring them from one basket to another under therapist supervision. Alongside VR, participants also underwent Routine Physical Therapy (RPT) three times per week for six weeks, each 40-minute session consisting of a warm-up with diaphragmatic breathing, stretching, strengthening and cool-down.
  Interventions: Device: artificial intelligence
- Proprioceptive Neuromuscular Facilitation (Active Comparator): Participants in this group received Proprioceptive Neuromuscular Facilitation (PNF) therapy in addition to Routine Physical Therapy (RPT). PNF was administered three times per week for six weeks, with each session lasting 30 minutes at a moderate intensity (RPE 11-13). Specific PNF techniques were selected for symptom management: slow reversal for kinetic tremor to improve coordinated agonist-antagonist contractions, rhythmic initiation for bradykinesia to facilitate movement initiation, and tactile input to enhance proprioception and body awareness. PNF was administered under the direct guidance of a physical therapist, with manual contact and graded resistance tailored to individual capacity. Participants also received RPT on the same schedule and with the same structure as described for the experimental group, including warm-up breathing, targeted stretching and strengthening, and cool-down static stretches.
  Interventions: Other: Intervention 1

INTERVENTIONS:
Other: Intervention 1 — Participants in the control group received Proprioceptive Neuromuscular Facilitation (PNF) therapy three times per week for a total duration of six weeks. Each session lasted approximately 30 minutes and was conducted at a moderate intensity, corresponding to an RPE of 11-13 on the Borg scale. For kinetic tremors, the slow reversal technique was applied. For bradykinesia, the rhythmic initiation technique was used. And to enhance proprioception, tactile input was provided through manual contact, resistance, and stretch applied by the therapist at key points of the movement pattern.
  Other Names: Proprioceptive Neuromuscular Facilitation
  Arms: Proprioceptive Neuromuscular Facilitation
Device: artificial intelligence — Participants in the experimental group underwent Virtual Reality (VR) training three times per week for a total of six weeks. Each session lasted approximately 30 minutes and was conducted at a moderate intensity, defined by the repetition of VR tasks five times per session. The intervention was delivered using the Oculus Meta Quest 2 head-mounted display, providing an immersive and interactive environment under the close supervision of a licensed physical therapist. The central activity involved 2 modules. Ball Shifting Module picking and placing five virtual balls within the simulated environment and transferring them from one basket to another. Cube Navigation Module, in this task, users guide a virtual cube through highlighted cells or routes using deliberate movements, requiring precise hand positioning and controlled movement paths.
  Arms: Virtual Reality

SUMMARY:
Parkinson's Disease is a chronic neurodegenerative disorder marked by the progressive loss of dopaminergic neurons in the substantia nigra and accumulation of α-synuclein (Lewy bodies).It impacts both motor and non-motor systems, with growing global prevalence-affecting 7-10 million people, mostly men over 60 years-due to increasing life expectancy and demographic shifts.

PD shows motor symptoms like tremors and bradykinesia, along with non-motor issues like depression, REM sleep disorder, and cognitive decline. Diagnosis is often delayed due to subtle early signs like constipation or shoulder pain and atypical cases lacking classical tremors.

VR offers immersive, task-specific therapy that enhances motor learning and neuroplasticity in a safe, engaging environment. By integrating sensory feedback and real-time motion tracking, VR reduces tremors, promotes cortical reorganization (notably in the sensorimotor cortex and cerebellum), and increases rehabilitation motivation through gamified experiences.

PNF is a hands-on therapy using tactile, auditory, and proprioceptive cues to improve coordination, strength, and movement patterns. Especially useful in Parkinson's rehabilitation, PNF targets rigidity, bradykinesia, tremors, and postural instability by reinforcing neuromuscular coordination and improving movement execution in functional, diagonal planes.

Sensorimotor control is the dynamic integration of sensory input, motor planning, and execution, which becomes disrupted in PD due to impaired proprioception and feedback loops. Patients rely excessively on visual feedback, making movement effortful, highlighting the need for focused upper limb rehabilitation strategies.

DETAILED DESCRIPTION:
* Experimental: (VR+ RPT) Participants in this group received Virtual Reality (VR)-based training in addition to Routine Physical Therapy (RPT). The VR intervention was delivered using the Oculus Meta Quest 3 headset and consisted of immersive, goal-directed tasks performed three times per week for six weeks, each session lasting 30 minutes at a moderate intensity (RPE 11-13). VR tasks were designed to target specific motor impairments, including pick-and-place tasks for kinetic tremor reduction, tracing tasks to address bradykinesia, and reaching and grasping tasks to improve proprioception. Participants interacted with five virtual balls in a simulated environment, transferring them from one basket to another under therapist supervision. Alongside VR, participants also underwent Routine Physical Therapy (RPT) three times per week for six weeks, each 40-minute session consisting of a warm-up with diaphragmatic breathing, 30 minutes of stretching and strengthening for the core, hip, knee, back, and elbow extensors, and a cool-down with static stretches for major muscle groups.
* Control: (PNF+RPT) Participants in this group received Proprioceptive Neuromuscular Facilitation (PNF) therapy in addition to Routine Physical Therapy (RPT). PNF was administered three times per week for six weeks, with each session lasting 30 minutes at a moderate intensity (RPE 11-13). Specific PNF techniques were selected for symptom management: slow reversal for kinetic tremor to improve coordinated agonist-antagonist contractions, rhythmic initiation for bradykinesia to facilitate movement initiation, and tactile input to enhance proprioception and body awareness. PNF was administered under the direct guidance of a physical therapist, with manual contact and graded resistance tailored to individual capacity. Participants also received RPT on the same schedule and with the same structure as described for the experimental group, including warm-up breathing, targeted stretching and strengthening, and cool-down static stretches.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's Disease according to Gelb's criteria
2. Stage II-IV Hoehn &Yahr scale
3. Intact cognition status (MMSE > 24)
4. 50-80 years of age

Exclusion Criteria:

1. History of PD surgery
2. Phobia of virtual gaming systems
3. Visual anomalies
4. Cardiovascular problems
5. Severe dyskinesia or "on-off" fluctuations

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Kinetic Tremors | 6 weeks
  Kinetic Tremors It is going to be measured by: Fahn-Tolosa-Marin tremor rating scale with internal consistency of Cronbach's α = 0.90.
  FTMTRS - Kinetic Tremor Section
  Rate the severity of tremor during each task using the following scale:
  1. Writing: _______
  2. Drawing (Archimedes spiral): _______
  3. Pouring water: _______
  4. Drinking from a cup: _______ • Total Kinetic Tremor Score: _______/16 (0 = No tremor, 1 = Mild, intermittent, 2 = Moderate, intermittent or mild, continuous, 3 = Marked, intermittent or moderate, continuous, 4 = Severe, continuous)
Bradykinesia | 6 weeks
  It is going to be measured by: MDS-UPDRS Part III with internal consistency of Cronbach's α: 0.90-0.93.
  MDS-UPDRS Part III - Bradykinesia Items (3.4-3.6)
  Rate each movement on a scale from 0 (normal) to 4 (severe):
  1. 3.4 L&R Finger Tapping: _______
  2. 3.5 L&R Hand Movements (open/close hands): _______
  3. 3.6 L&R Pronation-Supination of Hands: _______ • Total Bradykinesia Score (3.4-3.6): _______/24
Proprioception | 6 weeks
  •It is going to be measured by: Fugl Meyer UE Proprioception subscale with internal consistency of Cronbach's α: at 0.94-0.98.
  Scoring:
  0 = Only a few degrees (less than 10° in shoulder)
  1. = Decreased
  2. = Normal
  Shoulder Movement 0 1 2 Flexion (0°-180°) ☐ ☐ ☐ Abduction (0°-90°) ☐ ☐ ☐ External Rotation ☐ ☐ ☐ Internal Rotation ☐ ☐ ☐ Elbow Movement 0 1 2 Flexion ☐ ☐ ☐ Extension ☐ ☐ ☐ Forearm Movement 0 1 2 Pronation ☐ ☐ ☐ Supination ☐ ☐ ☐ Wrist Movement 0 1 2 Flexion ☐ ☐ ☐ Extension ☐ ☐ ☐ Fingers Movement 0 1 2 Flexion ☐ ☐ ☐ Extension ☐ ☐ ☐

CONTACTS AND LOCATIONS:
Overall Officials: Shoaib Waqas, PhD, Study Chair — Lahore University of Biological and Applied Sciences; Javeria Younas, DPT, Principal Investigator — Lahore College of Physical Therapy; Fatima Rehan, DPT, Principal Investigator — Lahore College of Physical Therapy; Laiba Dhillon, DPT, Principal Investigator — Lahore College of Physical Therapy
Locations (1):
- Lahore University of Biological and Applied Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
After the publication
Supporting Information: Study Protocol, SAP
Time Frame: June 2026- October 2026